CLINICAL TRIAL: NCT05974228
Title: Bioglass Wound Dressing in Treatment of Chronic Wound in Different Stage：a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Yunfeng Li (Unknown)
Responsible Party: Principal Investigator, Long Zhang, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2023-CW-Bioglass
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Chronic Wound
Keywords: Chronic wound; Bioactive glass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bioactive glass wound dressing — Bioactive glass wound dressing is a dressing covered on the wound bed

SUMMARY:
The goal of this randomized control trial is to test the efficacy and safety of a bioglass wound dressing in patients with chronic wound in different stages. The main question it aims to answer are:

* Whether the bioglass wound dressing have better efficacy and safety than blank control in treatment of chronic wound in necrosis stable stage？
* Whether the bioglass wound dressing have better efficacy and safety than blank control in treatment of chronic wound in granulation growth stage？ Participants will be assigned with a 1:1 ratio into intervention group and control group.

Participants of intervention group will receive bioglass wound dressing in addition with clinical optimal treatment plan. Participants of control group will only receive clinical optimal treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is aged 18-80 years old;
2. Ulcerative wounds;
3. In the stage of stable necrosis or granulation growth;
4. Voluntarily participate in this study and sign an informed consent form

Exclusion Criteria:

1. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, and respiratory failure have not been corrected yet;
2. Uncontrolled blood glucose, Glucose test#Fasting blood sugar>15mmol/L, Glycated hemoglobin>12%;
3. There is active bleeding inside the wound, and routine basic treatment plans cannot be implemented;
4. Serum albumin < 20 g/L; Hemoglobin<60 g/L; Platelets<50 × 10^9/L;
5. Spreading infection status, currently or about to be treated with antibiotics;
6. Patients with advanced malignant tumors;
7. Active period of autoimmune diseases;
8. Previous allergies to bioactive glass ointment dressings (self originating);
9. The patient is unable to cooperate or has mental disorders;
10. According to the judgment of the researcher, the subject has a clear reason that cannot be removed and affects wound healing, which is not suitable for this study or cannot comply with the requirements of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
2-week reduction rate of wound area | 2-week

SECONDARY OUTCOMES:
2-week wound healing rate | 2-week

IPD SHARING:
Plan to Share IPD: No